CLINICAL TRIAL: NCT05694039
Title: A Prospective Cohort Study On Change of Cognitive Function In Aged-related Hearing Loss With Hearing Aids
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SunYatsenU2H_YangH02
Record Dates: First submitted 2023-01-12; First posted 2023-01-23 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2022-03

CONDITIONS: Age-related Hearing Loss; Hearing Loss, Sensorineural; Hearing Aid; Cognitive Function Abnormal
MeSH Terms: conditions — Presbycusis; Hearing Loss, Sensorineural; Cognition Disorders | interventions — Hearing Aids

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Procedure: no intervention
- Intervention Group (Active Comparator): Procedure: a intervention via hearing aids for 5 years
  Interventions: Device: Hearing Aids

INTERVENTIONS:
Device: Hearing Aids — The intervention group uses hearing aids, and the intervention group receives hearing aid intervention for 5 years.
  Arms: Intervention Group

SUMMARY:
Background:

Deafness is one of the nine potentially modifiable risk factors for dementia simulated by the Lancet dementia Prevention, intervention and Care Committee in 2017. Some studies have found that the risk factors of dementia in deafness system, with the increase of the degree of deafness, the risk of cognitive decline increases, while after long-term wear of hearing aids, the deterioration of immediate and delayed memory is less, and the possibility of cognitive decline slows down. Therefore, it is necessary for us to improve the auditory ability of patients with deafness through auditory intervention, so as to slow down its effect on dementia and reduce the incidence of dementia. At present, auditory intervention methods include hearing aid wearing and cochlear implant.

However, there are few studies on cognitive function of presbycusis patients in China, and there is no research on how many years of auditory intervention can effectively slow down the incidence of dementia in presbycusis patients with MCI. Therefore, we intend to conduct a prospective cohort study on the changes of cognitive function of presbycusis under hearing aid intervention.

DETAILED DESCRIPTION:
Materials and methods: The unicentric, prospective cohort study included 388 patients with presbycusis aged 60-85 who were recruited in the Department of Otorhinolaryngology from March 2022 to March 2028. They were averagely divided into the control group (n = 194) and the intervention group (n = 194). The post intervention group received hearing aid intervention, and was followed up for 5 years, once every six months. Audiological assessment, cognitive function assessment, noninvasive brain imaging assessment and hearing aid effect assessment were performed at baseline and each follow-up. This thesis aim to investigate the changes of cognitive function in senile deafness under the intervention of hearing aids.

ELIGIBILITY:
Inclusion Criteria:

Age>60yrs，≤85yrs（MCI prevalence was 6.7% for ages 60-64, 8.4% for 65-69, 10.1% for 70-74, 14.8% for 75-79,and25.2% for80-84）; Sensorineural Hearing loss with pure-tone thresholds 25-70 dB HL at octave frequencies between 250 and 4000 Hz, 4 frequency PTA of ≥ 30 dB HL, and the PTA ≤ 90 dB HL; Diagnosed as Presbycusis; Score of 23 or below on Mini-Mental Status Exam (MMSE); Score of 22 or below on Montreal Cognitive Assessment (MoCA);

Exclusion Criteria:

Hearing loss exceeding the limits that can be successfully aided with hearing aids (i.e., profound hearing loss); Significant history of otologic or neurologic disorders; Hearing loss remediated with a cochlear implant (cannot wear hearing aids); Any clinically significant unstable or progressive medical condition; Any condition which, in the opinion of the investigator, places the participant at unacceptable risk if he or she were to participate in the study.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 388 (Estimated)
Dates: Start 2022-03-09 (Actual); Primary Completion 2028-03-09 (Estimated); Study Completion 2028-03-09 (Estimated)

PRIMARY OUTCOMES:
MoCA | half a year
  Montreal Cognitive Assessment is an assessment tool for rapid screening of cognitive dysfunction.
MMSE | half a year
  Mini-mental State Examination is currently the preferred scale for cognitive impairment screening and is widely used in dementia screening.

SECONDARY OUTCOMES:
Pure Tone Audiometry | half a year
  Pure audiometry is to measure the air conduction hearing thresholds of 125Hz, 250Hz, 500Hz, 1000Hz, 2000Hz, 4000Hz and 8000Hz and bone conduction threshold of 500Hz, 1000Hz, 2000Hz and 4000Hz in normal people and deaf patients by Hughson-Westlake(HW) method, also gets the tested person's pure-tone average (PTA) in the hearing ear which is calculated using thresholds for 0.5, 1, 2 and 4 kHz. The acoustic standard of the sound insulation room is GB/T16296, the reverberation time is (0.3±0.15) seconds, and the pure tone audiometer model is Interacoustics AC40(Inter-c AC40).
Speeeh Audlometry | half a year
  Speech audiometry is a kind of audiometry method that uses standardized speech signals as sound stimulation to test the speech recognition ability of subjects.

OTHER OUTCOMES:
EEG/ERP | half a year
  Electroencephalograph ( EEG power in alpha band) is record which reflects regular electric action of brain cells groups by the 128-channel EEG analyzer of EGI Company, USA, with its matching electrode cap, of which transverse axis represents time, and vertical y-axis represents value of potential generated by brain cells.
fNIRS | half a year
  Functional Near Infrared Spectroscopy uses fNIRS signal to measure the magnetic changes caused by the change of hemoglobin concentration in the process of brain cognitive activity at the level of brain imaging, so as to obtain BOLD signal.
Hearing Aid Assessment composite | half a year
  The assessment of hearing aid effect includes Chinese Version Hearing Handicap Inventory for the Elderly Screening(CHHIE-S), Abbreviated Profile of Hearing Aid Benefit(APHAB), Satisfaction with Amplification in DailyLife(SADL) and International Outcome Items for Hearing Aids(IOI-HA).

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China